CLINICAL TRIAL: NCT05383547
Title: Prospective Observation of Bortezomib in the Treatment of Glomerular Diseases
Brief Title: Bortezomib for Treating Glomerular Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Nan Chen,MD, Principal Investigator,Director,Foreign academicians of the French National Academy of Medical Sciences,Director of institute of Nephrology affiliated to Shanghai Jiao Tong University Medical College, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-53
Record Dates: First submitted 2022-05-10; First posted 2022-05-20 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-05

CONDITIONS: Bortezomib; Glomerulonephritis; MN; MPGN; FSGS; IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis; Glomerulonephritis, IGA | interventions — Bortezomib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glomerular disease patients (Experimental)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Dexamethasone 10mg+ bortezomib (1.3mg /m2 IV) was administered at D1,D4,D8,D11, one month for 1 cycle, for 2 cycles.

SUMMARY:
Bortezomib is a proteasome inhibitor that inhibits autoantibody production, and reduces podocyte damage and mesangial hyperplasia caused by NF-κB activation in the kidney. Literature has reported that bortezomib can achieve a complete response rate of up to 38% in the treatment of glomerular diseases, but its safety and effectiveness remain to be assessed for the Chinese demographic. This study attempts to explore a new treatment plan for glomerular disease by observing the therapeutic effect of bortezomib on glomerular disease.

ELIGIBILITY:
Inclusion Criteria:

* Glomerular diseases confirmed by renal biopsy (including IgA nephropathy, membranous nephropathy, FSGS, etc.)
* Aged 18-65, male or female
* Signed informed consent
* 24h proteinuria >1.5g/24h
* Glomerular filtration rate (eGFR) >30ml/min/1.73m2 (calculated according to CKD-EPI formula) within 14 days before enrollment.
* Blood pressure <140/90mmHg after drug treatment
* Unless there are contraindications, subjects must take a steady dose of ACEI and/or ARB for at least 4 weeks before screening

Exclusion Criteria:

* Renal pathology: glomerulosclerosis ratio >70%, interstitial fibrosis > severe
* Received immunosuppressant treatment within the past 6 months
* Inability to tolerate bortezomib
* Platelet count < 30×109/L within 14 days before enrollment
* Neutrophil count < 1.0×109/L within 14 days before enrollment
* Subjects had >grade 2 peripheral neuropathy within 14 days before enrollment
* ECG evidence of myocardial infarction or NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmia, or acute ischemia or active conduction system abnormalities within 6 months before enrollment
* Abnormal liver function such as alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >=3 times normal upper limit (ULN), total bilirubin >= 2 times ULN
* Newly diagnosed malignant tumor (within 5 years) or undergoing radiotherapy/chemotherapy
* Women who are pregnant or breast-feeding, or women of childbearing age who cannot guarantee effective contraception
* New serious life-threatening infections
* Active infectious diseases such as active tuberculosis, active viral hepatitis, HIV infection.
* Mental disorders and psychotropic drug uses
* Patients with an estimated life expectancy of fewer than 12 months
* Patients that were difficult to follow up on or had poor compliance
* Patients who do not wish to sign the form of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate of Proteinuria | One Year
  24h Proteinuria <300mg/24h

SECONDARY OUTCOMES:
Safety of Bortezomib | One Year
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China